CLINICAL TRIAL: NCT06643429
Title: Impact of Environmental Factors and Metabolomics on Colorectal Cancer Development and Prognosis Based on Environmental Factors and Metabolomics.
Brief Title: Impact of Environmental Factors and Metabolomics on Colorectal Cancer.
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2024-222-02
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Metabolic Disease
Keywords: colorectal cancer; air pollution; metabolomics; intestinal flora
MeSH Terms: conditions — Colorectal Neoplasms; Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- the control group: Adults with no history of malignancy and willing to participate in this study.
- the colorectal cancer group: Patients with preoperative diagnosis of colorectal cancer confirmed by pathological biopsy.
  Interventions: Diagnostic Test: colorectal cancer
- the colorectal adenoma group: Patients with preoperative diagnosis of colorectal adenoma confirmed by colonoscopy.
  Interventions: Diagnostic Test: colorectal neoplasm

INTERVENTIONS:
Diagnostic Test: colorectal cancer — Patients diagnosed with colorectal cancer by pathological biopsy.
  Groups: the colorectal cancer group
Diagnostic Test: colorectal neoplasm — Patients diagnosed with colorectal adenoma confirmed by colonoscopy.
  Groups: the colorectal adenoma group

SUMMARY:
Colorectal cancer is one of the malignant tumours with high morbidity and mortality worldwide, posing a serious threat to human health. In recent years, the incidence of colorectal cancer has been on the rise with changes in lifestyle and dietary habits. Although some progress has been made in treatments such as surgery, chemotherapy and radiotherapy, however, the early diagnosis, prognosis assessment and personalised treatment of colorectal cancer still face great challenges. Therefore, it is of great academic value and practical significance to deeply explore the influencing factors of colorectal cancer occurrence, development and its prognosis, especially the research on environmental factors and metabolomics.

DETAILED DESCRIPTION:
In this study, investigators collected clinical information, blood, urine and stool for ambient air pollution analysis, blood metabolomics analysis and stool macro-genetic sequencing by including patients from healthy control and colorectal cancer groups, respectively. Environmental factors, metabolomics and intestinal microbiota data were integrated and analysed to screen for indicators that play a key role in colorectal cancer development and construct a colorectal cancer prediction model.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy control group:

   * age ≥18 years old;
   * no history of malignant tumour;
   * willing to participate in this study and sign the informed consent form;
   * complete basic data.
2. Gastric cancer group:

   * age ≥18 years old;
   * patients diagnosed with gastric cancer by pathological biopsy before operation;
   * no chemotherapy, radiotherapy, targeted and immunotherapy before enrolment;
   * willing to participate in this study and sign the informed consent; complete clinical data.

Exclusion criteria:

* patients with primary malignant tumours other than gastric cancer;
* patients with serious cardiopulmonary insufficiency and other systemic diseases that affect the choice of treatment plan;
* patients who are not suitable for enrolment as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients diagnosed with colorectal cancer and undergoing radical surgery for colorectal cancer at the study centre.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative complications | From date of surgery until the date of first documented postoperative complication, assessed up to 2 months after surgery.
  Surgical complications was defined as any postoperative complication occurring during the postoperative hospitalisation period.

SECONDARY OUTCOMES:
Overall survival | From date of diagnosis until the date of death from any cause or or loss to follow-up, whichever came first, assessed up to 60 months.
  Overall survival was defined as time from date of diagnosis until the date of death from any cause or or loss to follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No